CLINICAL TRIAL: NCT06127771
Title: Examining the Effects of Unblocking the Full Potential of Medtronic PerceptTM PC IPG on Symptoms of Individuals with Parkinson's Disease
Brief Title: Effects of Unblocking the Full Potential of Percept PC IPG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Alfonso Fasano, Dr. Alfonso Fasano, MD, PhD, FAAN, Professor, Department of Medicine, Division of Neurology at University of Toronto, Toronto Western Hospital, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 23-5697
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care programming (No Intervention): Individuals' DBS will be programmed using SOC programming parameters.
- Percept PC programming (Experimental): Individuals' DBS will be programmed using the full capacity of Percept PC IPG.
  Interventions: Other: Programming DBS using Percept PC neurostimulator's full potential

INTERVENTIONS:
Other: Programming DBS using Percept PC neurostimulator's full potential — This study aims to enroll patients who previously had Activa PC neurostimulator and underwent a battery change to Medtronic PerceptTM PC as standard-of-care. However, in this study, the investigators intent to fully utilize the programming potential of Medtronic PerceptTM PC to optimize treatment outcome.
  Arms: Percept PC programming

SUMMARY:
Population Size and Eligible Patients: The study will enroll patients with Parkinson's disease (n=30) who had an IPG replacement from Activa PC (older generation of neurostimulator) to Medtronic PerceptTM PC (newer generation of neurostimulator) as a part of their standard-of-care. No patient will be receiving the system for research purposes only.

Study Design: This is a prospective, double-blinded, randomized, cross-over clinical investigation to further investigate the efficiency of Medtronic PerceptTM PC neurostimulator. This study involves three in clinic visits. During the first study visit, the patients' neurostimulator will be reprogrammed using all the additional features the Percept PC has to offer. At the end of the visit, the patients will be randomized between their baseline program, ((Activa PC group) and the newly defined programming settings (Percept Group). During the second visit (1-month follow-up) the effect will be clinically assessed, and a crossover of the condition will happen. The third visit (2-month follow-up) will be a follow-up visit with no programming but only clinical assessment.

Study Duration: Expected study duration is 1 year with the possibility for renewals.

Objectives and outcome measures: The goal is the study is to define whether or what the benefit is of the Percept PC neurostimulator compared to the older Activa PC neurostimulator. The primary outcome is patient-reported global impression of change (PGIC). The secondary outcome measures are clinical scales assessing symptoms of Parkinson's disease (UPDRS-III and -IV) and quality of life (PDQ-39), the active problems list and amount of medication intake.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with idiopathic Parkinson's disease who previously underwent DBS surgery.
* Individuals who had IPG replacement from Activa PC to Medtronic PerceptTM PC Neurostimulator as standard-of-care
* Individuals should be able to provide their informed consent

Exclusion Criteria:

* Cognition impairment (MoCA < 20/30)
* Patients with severe PD symptoms who are unable to come to the clinic three times within three months (e.g. bedridden patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-09-29 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Patients' Global Impression of Change (PGIC) scale | First programming (Baseline) - Crossover programming (1 month Follow-up)- Third month Follow-up
  the investigators expect to see an improvement of PGIC due to a decrease in (the severity of) active problems. The PGIC scale ranges from 1 to 7, with 1 indicating no change and 7 signifying a substantial improvement.

SECONDARY OUTCOMES:
MDS-UPDRS-III | First programming (Baseline) - Crossover programming (1 month Follow-up)- Third month Follow-up
  the investigators expect to see an improvement in the MDS-UPDRS-III. Part III: Motor examination: 0 to 132, with higher scores indicating greater motor impairment.
MDS-UPDRS-IV | First programming (Baseline) - Crossover programming (1 month Follow-up)- Third month Follow-up
  the investigators expect to see an improvement in the MDS-UPDRS-IV. The score ranges from 0-24. Higher scores indicate more severe impairment.
The Parkinson's Disease Questionnaire (PDQ-39) | First programming (Baseline) - Crossover programming (1 month Follow-up)- Third month Follow-up
  the investigators expect to see an improvement in PDQ-39. 0 to 100; being the higher the score, the worse the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Movement Disorders Centre - Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No